CLINICAL TRIAL: NCT03911726
Title: Do Antipsychotic Agents Induce Supersensitivity in Humans: A Combined PET/MRI Study in Patients With Schizophrenia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-09-18
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia
Keywords: PET/MR; Dopaminergic supersensitivity; D2/3 receptor availability
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: All study participants will undergo a single PET/MR-measurement.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy subjects (Other): 30 healthy subjects will undergo a single PET/MR-measurement.
  Interventions: Radiation: Single PET/MR-measurement
- First-episode, drug-naive patients with schizophrenia (Experimental): 20 first-episode, drug-naive patients with schizophrenia will undergo a single PET/MR-measurement.
  Interventions: Radiation: Single PET/MR-measurement
- Pretreated chronically ill patients with schizophrenia (Experimental): 90 pretreated chronically ill patients with schizophrenia will undergo a single PET/MR-measurement.
  Interventions: Radiation: Single PET/MR-measurement

INTERVENTIONS:
Radiation: Single PET/MR-measurement — A single PET/MR-measurement using [18F]Fallypride with a duration of 180min. Within this measurement, the dopamine receptor agonist apomorphine is applicated.

SUMMARY:
The aim of the present study is to detect changes in the dopamine system in the brain of patients with schizophrenia, especially when pretreated with antipsychotic medication. Here, the investigators want to find out whether the treatment with these drugs can cause permanent changes in docking points (receptors) of dopamine in the brain. It will be examined whether number and response of dopamine receptors is altered, which are associated with the onset of psychotic symptoms. For this purpose, a single PET/MR measurement will be performed in all participants. In total 140 volunteers, consisting of 30 healthy volunteers, 20 first-episode, drug-naive patients with schizophrenia and 90 pretreated patients with schizophrenia will be included over a time period of three years. In addition, the influence of nicotine consumption on dopamine receptors will be invesitgated by comparing data from smoking and non-smoking patients. In clinical practice, an elevation of dopamine action caused by alterations in receptors in the brain is of most importance. This may be the reason why the treatment with antipsychotic agents does not work in some patients. In addition, a permanent elevation of dopamine action is associated with permanent brain alterations by these drugs. The result can contribute to work out valuable indications, whether it makes sense to continue a long term therapy with antipsychotic drugs in a patient. But also the in-depth understanding of the impact of nicotine on the course of therapy can help to open up possibilities for improved drug treatment.

DETAILED DESCRIPTION:
This project will study for the first time in humans, whether long-term treatment with antipsychotic agents, representing nowadays gold standard for patients with schizophrenia, may lead to an up regulation of dopamine D2-like receptors and associated, a supersensitivity of these receptors. The detection of such changes and the study of influencing factors (in particular smoking and type of medication) are most important for the understanding of relapse risks, development of treatment resistance and the risks for motor complications of antipsychotic pharmacotherapy. This monocentric, controlled study will include 140 participants over a time period of three years. 30 healthy volunteers, 20 first-episode, drug-naive patients with schizophrenia and 90 pretreated patients with schizophrenia will undergo a single PET/MR measurement.

ELIGIBILITY:
Inclusion Criteria for healthy subjects:

* Age: 18-65
* The subject is capable to understand scope and individual consequences of the clinical study.
* An informed consent is signed and personally dated by the subject. • No psychiatric disorder (DSM-5) currently, or in the medical history (ensured by a standardized psychiatric interview Mini International Neuropsychiatric Interview (M.I.N.I.)).

Inclusion Criteria for patients:

* Age: 18-65
* The criteria for schizophrenia after DSM-5 are met.
* The subject is capable to understand scope and individual consequences of the clinical study.
* For first-episode patients, no application of antipsychotic drugs in history. Other psychoactive substances (in particular antidepressants) are allowed if last application is at least three months ago and total Duration did not exceed three months. Benzodiazepines are allowed.
* For medically pretreated patients: at least one year pharmacotherapy with one of the following three substances: aripiprazole or quetiapine or risperidone. A medication break of - depending on the plasma level - two days (quetiapine) up to two weeks (aripiprazole) should be clinically defensible.
* An informed consent is signed and personally dated by the patient. For patients with legal support in addition: signature of the legal supervisor.

Exclusion criteria for patients and subjects:

* Hypersensitivity against apomorphine or a chemically similar substance or one of the components of the applied medication.
* Participation in other clinical trials during or within six months prior to this clinical study.
* Medical or psychological conditions which may endanger a proper performance of the clinical trial.
* Physical disorders which interfere according to type and severity with the planned examinations, which could influence the parameter to be investigated or could compromise the subject during the examination procedure.
* Inability to comply with the study protocol.
* Limited or completely repealed legal capacity.
* For female participants: positive pregnancy test on the day of the study inclusion or on the day of the PET/MR-measurement.
* Acute suicidality or endangerment
* Poor general condition.
* Participation in a study using ionising Radiation within the last five years.
* Alcohol abuse, alcohol dependence or addiction disease / abuse of dependence-inducing substances (excluding nicotine) in the history, additional exclusion criterion for healthy subjects: regular medication intake; within the last two weeks before PET/MR-measurement no drugs at all must be taken.

Additional exclusion criterion for patients: other than the approved axis I diagnosis according to DSM-5. An axis II diagnosis is not a criterion for exclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Dopamine D2/D3-receptor availability | 160 minutes
  Dopamine D2/D3-receptor availability measured as binding potential (BP) using PET and blood-oxygen-level-dependant (BOLD)-response measured with fMRI.

SECONDARY OUTCOMES:
D2/D3-receptor availability in first-episode, drug-naive patients with schizophrenia | 160 minutes
  In first-episode, drug-naive patients with schizophrenia expressions of NSS and AIMS correlate significantly with striatal D2/D3-receptor availability.
D2/D3-receptor availability in patients with TD | 160 minutes
  In pretreated, chronically ill patients with schizophrenia, patients with TD show a significantly higher D2/D3-receptor availability than patients without TD.
Follow-up of pretreated, chronically ill patients with schizophrenia | two years
  In pretreated, chronically ill patients with schizophrenia, the D2/D3-receptor availability correlates with the relapse risk and the risk for the development of TD over the course of two years.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Gründer, Prof. Dr., Principal Investigator — Central Institute of Mental Health, Mannheim
Locations (1):
- Central Institute of Mental Health, Mannheim, Baden-Wurttemberg, Germany